CLINICAL TRIAL: NCT04255745
Title: The Impact of a Resistance Training Intervention on Blood Pressure Control in Older Adults With Sarcopenia
Acronym: INERTIA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Deepika Laddu-Patel, Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-0009; 1K01HL148503-01 (NIH)
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Sarcopenia; High Blood Pressure; Hypertension
Keywords: cardiovascular disease prevention; aging; exercise; blood pressure; sarcopenia; resistance training; older adults
MeSH Terms: conditions — Sarcopenia; Hypertension; Motor Activity

STUDY DESIGN:
Intervention Model Description: permuted block randomization scheme,
Who Masked: Investigator
Masking Description: Primary investigator will be masked to the outcome data collection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Assessment-only control (No Intervention): 30 Assessment-only control group will be mailed (standard or electronic) NIH/National Institutes on Aging (NIA) Go4Life® educational materials once a month for 3 months. Exercise logs documenting weekly exercise activities, duration, time and effort will be requested to be sent back.
- Intervention (Experimental): 60 Intervention group will receive 12 weeks of supervised resistance training following the American Heart Association and American College of Sports Medicine guidelines for older adults. Exercises will include a mixture of upper-body and lower body strength exercises. Training load will be determined based on initial 1-repetition maximum tests (1-RM). Initial exercise load will start off at low resistance (40-50% 1RM) with more frequent repetitions per exercise, and will gradually increase weight load and intensity over the exercise training period.
  Interventions: Behavioral: progressive resistance training

INTERVENTIONS:
Behavioral: progressive resistance training — Individual, tailored, progressive muscle strength and function intervention
  Arms: Intervention

SUMMARY:
Current prevention and treatment of high blood pressure (BP) in sarcopenia, by non-pharmacological approaches remain limited and are far from optimal. This randomized control intervention pilot study will provide new evidence of the unexplored relationship between muscle strength and high BP in sarcopenia, and experimentally test the effects of an evidence-based progressive resistance training intervention on BP, while also examining reversibility to identify muscle strength as a non-pharmacological target for BP control in older sarcopenic adults.

DETAILED DESCRIPTION:
This premise of this K01 proposal is to address current gaps in the literature regarding the understanding of high blood pressure due to sarcopenia, and provide new evidence for the discernible relationship between low muscle strength and blood pressure in sarcopenia, and effective non-pharmaceutical treatment approaches. This study will evaluate the feasibility of recruitment, retention, implementation and adherence to an empirically-based progressive resistance training (PRT) intervention to test its effect on blood pressure in a targeted population of older adults with sarcopenia who are randomized (via block permuted scheme) to the PRT intervention. Built within this randomized control intervention design, the investigators will further explore reversibility to examine whether muscle strength serves as an intervention target for blood pressure control in sarcopenic adults, which will be more appropriately tested in subsequently well-powered R-level intervention studies. Physiologically plausible microvascular mechanisms by which the PRT impacts changes in blood pressure will also be explored.

ELIGIBILITY:
Inclusion Criteria:

* Adults (men and women) aged 60 years and older (any racial/ethnic background)
* Demonstrates adequate cognitive function by the MoCA (education adjusted score of >22 at screening)
* Sedentary or low active adults (not active in strength training)
* Resides in the Chicagoland Area
* Able to walk/perform exercise without complete dependence on assisted device
* Able and willing to enroll and provide written informed consent, i.e., to meet the time and data collection requirements of the study, be randomized to 1 of 2 treatment arms, follow through assignment during 3 months active period, participate in 1 follow-up visit at 12 months

Exclusion Criteria:

* Subjects with self-report of inability to walk at least ¼ mile or walk 400 meters in <15 minutes without sitting
* Subjects who self-reported having a history of a cardiovascular disease event or physician diagnosed cardiovascular disease (heart attack, heart failure, congenital heart disease, peripheral vascular disease, coronary revascularization, or angina that required overnight hospitalization), cerebrovascular disease (stroke, transient ischemic attack)
* Diagnosis of cancer (other than non-melanoma skin cancer) that is/was active or treated with radiation or chemotherapy within the past 5 years;
* Subjects with orthopedic pathology or deformity that prevents exercising safely
* Diagnosis or history of cognitive impairment (Dementia, Alzheimer's Disease) or bipolar or psychotic disorder or hospitalization for psychological or emotional problems within the last 2 years
* Diagnosis of autoimmune diseases, such as (but not limited to) lupus, multiple sclerosis, advanced/severe rheumatoid arthritis that would preclude exercising safely
* Diagnosis of advanced or severe osteoporosis or orthopedic deformities that may prevent strength training exercise safely
* Participants from the same household as those already enrolled in the study
* Current abuser of alcohol or usage of illicit drugs or history of alcohol or drug abuse
* Planning to move out of the area or take an extended vacation during the study period
* Current or planned participation in in another structured program that overtly focuses on exercise
* Currently enrolled or planning to enroll into another research study that would limit full participation in the study
* Investigator discretion for clinical safety or protocol adherence reasons

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2020-01-27 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2025-05-01 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure | baseline, 12 weeks, 1 year
  change in systolic and diastolic blood pressure

SECONDARY OUTCOMES:
Short Physical Performance Battery (SPPB) | baseline, 12 weeks, 1 year
  4 meter gait speed (m/s; slow speed indicates lower function), timed five-time-sit-to-stand (in seconds, slower time indicates lower function), 3-stage balance (3 positions total, scored separately; inability to hold each position for 10seconds each indicates lower function)
Timed up and go performance | baseline, 12 weeks, 1 year
  change in timed up and go (slower time indicates lower function)

OTHER OUTCOMES:
Muscle strength | baseline, 8 weeks 12 weeks, 1 year
  muscle strength will be assessed using the 1 Repetition maximum test ( the maximum amount of weight a person can hold while performing an exercise safely and maintaining form. the 1RM will be tested on upper and lower body for a total of 6 exercises, as recommended by the American College of Sports Medicine. Changes in 1RM will be reevaluated to see if strength improves.
  1. chest press
  2. leg press
  3. lat-pull down
  4. leg extensions
  5. shoulder press
  6. leg curls
Microvascular flow-induced vasodilation (FID) dose response | baseline, 12 weeks
  Microvessels in subcutaneous fat (SF) will be extracted from 10 intervention and 5 control subjects (total=15) and isolated for microvascular flow-induced vasodilation (FID). Microvessels will be constricted to physiological and pharmacological pressures (stimuli) followed by dialation by a vasodialtor. The dose response curves to vasodialator will be measured (known as FID dose-response) will be the primary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Deepika Laddu, PhD, Principal Investigator — Northwestern University
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Laddu D, Kim H, Phillips SA, Ma J. INERTIA: A pilot study of the impact of progressive resistance training on blood pressure control in older adults with sarcopenia. Contemp Clin Trials. 2021 Sep;108:106516. doi: 10.1016/j.cct.2021.106516. Epub 2021 Jul 24. PMID 34311098